CLINICAL TRIAL: NCT07143981
Title: Fecal Microbiome Transplant to Normalize Gut Microbiota, Metabolomics, Immunology, Cognitive and Affective Processing in Patients Suffering From Anorexia Nervosa
Brief Title: The Fecal Microbiome Transplant (FMT) Study for Anorexia Nervosa
Status: Recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Western University, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: ANFMT-001
Record Dates: First submitted 2025-06-30; First posted 2025-08-27 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Anorexia Nervosa
Keywords: Microbiome; Fecal transplant; Gut microbiome; Gut brain axis; Mental health; Eating Disorders
MeSH Terms: conditions — Anorexia Nervosa; Psychological Well-Being; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Active treatment: Receiving FMT

SUMMARY:
Anorexia Nervosa (AN) is a severe, debilitating and potentially life threatening illness that is difficult to treat. A cardinal symptom of AN is the mistaken belief on the part of the individuals that they are overweight and must continue to restrict intake. This fixed false belief is a detrimental factor to recovery. It is known that AN involves disturbance in the gut microbiome (GM; the microbes that live in the lower intestinal tract). The GM also affects how one thinks and makes food choices - there appears to be a direct link between the GM and how the brain functions. This connection is thought to occur through chemical processes that convey information from the gut to the brain. It is known that fecal microbiome transplant (FMT) has been useful in treating several illnesses, including several mental illnesses. The investigators intend to deliver FMT to individuals with AN to determine the extent to which this modifies their GM, their biochemistry, their thinking processes and their moods and emotions. The investigators believe this will illuminate important aspects of AN that keep the illness in place, and that this will uncover useful approaches to better treat it.

DETAILED DESCRIPTION:
The overall objective is to determine FMT's acceptability and the extent and means by which it helps patients with AN, restricting type. The investigators hypothesize that FMT will lead to diversification of the GM, improved metabolic and immunological status and reduced cognitive and psychiatric symptoms in patients with AN, details never investigated before. This will be due to FMT's ability to impart healthy microorganisms into the lower intestines and, thereby, improve GBM-axis signaling that may contribute to maintaining AN. The investigators propose that this will result in measurable improvement in cognitive distortions about weight, leading to reduced AN symptomatology, breaking the weight loss/AN cycle.

Specific Aims & Hypotheses

This is a one-group, pre-/post-intervention trial of FMT in AN-restricting type, with 1-week, 3-week and 3-month follow up, administered before specialized eating disorders treatment. The hypotheses are:

1. FMT will result in a sustained increase diversity of microbes with the metabolomic characteristics of increased short-chain fatty acids and bacteriophage composition compared with pre-treatment, as determined by targeted metabolomic approaches.
2. FMT will improve immune profiles, reducing IL6, IL1b and the proportion of Th17 cells, along with an increase in repair cytokines such as TARC, IL4, IL13 and BDNF and Th2 cells.
3. FMT will significantly improve cognitive and affective functioning, including task-switching efficiency, food aversion and obsessional thinking about weight, punishment and reward sensitivity, depression and anxiety symptomatology, and AN symptom severity.

This is a prospective, longitudinal, single-arm, pre-post intervention. Variables will be compared using repeated-measures analyses with each participant as their own comparator.

ELIGIBILITY:
Inclusion Criteria:

* meet DSM 5 criteria for AN, restricting type, moderate or higher severity, as indicated by a BMI<17
* Participants must we willing and able to swallow FMT capsules without vomiting
* Able to read and understand conversational English

Exclusion Criteria:

1. Medical or psychiatric instability needing hospitalization
2. Patients with AN binge/purge type
3. Use of antibiotics or probiotics in the month prior to treatment
4. Regular oral steroid use, or potent topical steroid use on large sections of skin
5. Chronic immune compromise and chronic illness affecting the intestinal tract or metabolic health
6. Pregnancy or intended pregnancy over the time of study
7. Patients enrolled in any treatment program that involves refeeding

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants in this study will be awaiting treatment for anorexia nervosa at London Health Sciences Centre's (LHSC, Ontario Canada) Adult Eating Disorders Service (AEDS).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention | 1, 3, and 12 weeks post intervention
  Success will be evaluated using recruitment and retention rates, adverse event rates, and missing data rates. Scores at 75% or above will indicate high tolerability for this population that is in desperate need of additional intervention options.

SECONDARY OUTCOMES:
Shannon's Diversity Index | Pre-intervention, 12 weeks post-intervention
  Metric of microbiome diversity that considers richness of number of species and abundance. Higher values indicate more diversity. A value of 0 indicates that a community only has one species.
Activated blood cells producing Th17/Th2 cytokines | Pre-intervention, and 12-weeks post intervention
  Activated blood cells producing Th17/Th2 cytokines by Luminex - IL6, IL1b, IL17, IL4, IL13 to evaluate immune responses.
Activated blood cells producing BDNF | Pre-intervention and 12-weeks post-intervention
  Activated blood cells producing BDNF measured by Enzyme-Linked Immunosorbent Assay (ELISA)
RNA levels | Pre-intervention and 12-weeks post-intervention
  RT-PCR (reverse transcription-polymerase chain reaction) for RNA levels of CCR6, CRTh2, CCR4, CXCR5 (marker genes for Th17 and Th2 cells)
Task-switching Efficiency | Pre-intervention, and 12 weeks post-intervention
  -Task-switching efficiency measured using the Cued Color-Shape Switching Task, CCSST. Accuracy and response time will be computed on both single-task blocks and mixed task blocks, where participants will need to switch between colour and shape responses. Switch costs and mixing costs will be calculated from these scores.
Punishment sensitivity and reward sensitivity | Pre-intervention and 12-weeks post-intervention
  Punishment sensitivity and reward sensitivity using the Behavioural Inhibition System/Behavioural Activation System Scales (BIS/BAS). There are three BAS scales in which higher scores equate to greater sensitivity to reward. There is one BIS scale for which higher scores equate to greater sensitivity to punishment.
Depression | Pre-intervention, and at 1-, 3-, 12-weeks post intervention
  Depression evaluated using the Montgomery Asberg Depression Rating Scale (MADRS). It is a 9-item scale where higher score indicates more severe depressive symptoms.
Depression | Pre-intervention, and at 1-, 3-, 12-weeks post intervention
  Depression assessed with the Patient Health Questionnaire (PHQ-9), a 9-item scale evaluating the severity of depressive symptoms. Higher scores indicate more severe symptomatology.
Anxiety | Pre-intervention, and at 1-, 3-, 12-weeks post intervention
  Anxiety assessed using the Spielberger State/Trait Anxiety Inventory (STAI)
Anxiety | Pre-intervention, and at 1-, 3-, 12-weeks post intervention
  Anxiety assessed by the Generalized Anxiety Disorder 7-item scale (GAD-7)
Eating Attitudes | Pre-intervention, and 1-, 3-, 12-weeks post intervention
  -Food aversion and obsessional thinking about weight using the Eating Attitudes Test (EAT-26)
Anorexia Nervosa Symptoms | Pre-intervention, and at 1-, 3-, 12-weeks post intervention
  AN symptom severity with the Eating Disorders Examination Questionnaire (EDE-Q)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Osuch, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Research Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
This is a small feasibility study. While we would not make personally identifiable information public, even the basic demographic information could be used to re-identify a participant. In light of the nature of this study we do not feel it is in the interest of our participants to share data on a repository.

REFERENCES:
- See also: Provides theoretical support for this project — https://pubmed.ncbi.nlm.nih.gov/35743087/
- See also: Provides theoretical support for this project — https://pubmed.ncbi.nlm.nih.gov/38505265/